CLINICAL TRIAL: NCT01503580
Title: Studies of Psychiatric Predisposing Factors, Treatment-related Cardiovascular Effects, and Prognostic Factors Associated With Antimuscarinic Drug (Tolterodine) for Female Overactive Bladder Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 200712062M
Record Dates: First submitted 2011-09-24; First posted 2012-01-04 (Estimated); Last update posted 2013-10-31 (Estimated); Status verified 2013-10

CONDITIONS: Antimuscarinic Drug
MeSH Terms: interventions — Tolterodine Tartrate; Solifenacin Succinate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- antimuscarinic drug (Experimental)
  Interventions: Drug: tolterodine, solifenacin

INTERVENTIONS:
Drug: tolterodine, solifenacin — The enrolled women before March 2009 were treated with tolterodine 4 mg slow-release, and after March 2009 were treated with solifenacin 5 mg once a day for 12 weeks.

SUMMARY:
Overactive bladder syndrome (OAB) affects around 17 % of female population. However, the etiology of OAB was complicated and unclear in many aspects. In particular, the research about psychiatric aspect of etiology in OAB was paucity. Besides, research about prognostic factors and impact of cardiovascular system of OAB treatment was also paucity. Therefore the aims of the investigators study were (1) to analyze the etiology of OAB in psychiatric aspects; (2) to analyze the prognostic factors associated with tolterodine treatment; (3) to analyze the differences of cardiac conduction and heart rate variability before and after tolterodine treatment; (4) to analyze the differences of arterial stiffness between non-OAB and OAB female patients, and before and after tolterodine treatment.

ELIGIBILITY:
Inclusion Criteria:

* all cases are female patients with lower urinary tract symptoms

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 155 (Actual)
Dates: Start 2008-08; Primary Completion 2010-07 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Changes of heart rate variability after antimuscarinics | 3 months
  Changes of heart rate variability after 3-months' antimuscarinics treatment

SECONDARY OUTCOMES:
Changes of arterial stiffness after antimuscarinics treatment | 3 months
  Changes of arterial stiffness after 3-months antimuscarinics' treatment
Changes of psychologic distress after antimuscarinics treatment | 3 months
  Changes of psychologic distress after 3-months' antimuscarinics treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Gynecology,National Taiwan University Hospital, Taipei, Taiwan